CLINICAL TRIAL: NCT00931749
Title: The Effects of Low Intensity Ultrasound on Medial Tibial Cartilage Morphology in Patients With Mild or Moderate Knee Osteoarthritis: A Double Blind, Randomized Placebo-controlled Study.
Brief Title: Effects of Ultrasound Therapy on Cartilage Healing in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Adalberto Loyola-Sanchez/ MSc on Rehabilitation Sciences candidate, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIUSKOA-09-218
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Knee Osteoarthritis
Keywords: ultrasound therapy; knee cartilage thickness; knee cartilage volume; mild knee osteoarthritis; moderate knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low intensity Ultrasound group (Experimental)
  Interventions: Device: Low intensity pulsed ultrasound therapy
- Sham ultrasound group (Sham Comparator)
  Interventions: Device: Sham Low intensity pulsed ultrasound therapy

INTERVENTIONS:
Device: Low intensity pulsed ultrasound therapy — 1 MHz, Spatial Average Intensity of 0.2 W /cm2, pulsed duty cycle 20%, 9.5 minutes, Therapeutic dose= 112.5 J/cm2. Fixed application on the medial side of the knee joint. Three sessions per week, during 2 months ( 24 sessions)
  Other Names: Ultrasound Unit. Intelect Mobile, Chattanooga Inc.
  Arms: Low intensity Ultrasound group
Device: Sham Low intensity pulsed ultrasound therapy — The Ultrasound device will not have the transducer´s crystal, so no ultrasonic energy will be provided.
  Other Names: Ultrasound Unit. Intelect Mobile, Chattanooga Inc.
  Arms: Sham ultrasound group

SUMMARY:
The purpose of this study is to determine the effects of low intensity ultrasound therapy over the cartilage morphology (thickness and volume) of patients with mild or moderate knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) negatively influences the healthy aging process of the population. Until today, there are no interventions that have proved effective for enhancing the cartilage regeneration of these patients. The use of Low Intensity Ultrasound (LIUS) therapy has demonstrated promising effects on cartilage regeneration in vitro and in vivo. The aim of this study was to assess the effects of 24 sessions of LIUS on the cartilage volume and thickness of patients with grades 1 and 2 (medial joint space narrowing OARSI atlas 2007) knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 45 years old.
* Fulfillment of the clinical / radiological diagnostic criteria proposed by Altman, et al. for knee osteoarthritis.
* Medial Tibiofemoral Compartment joint space narrowing grades 1 OR 2 according to the OARSI atlas guide.
* Ability to read and understand English questionnaires and follow instructions.

Exclusion Criteria:

* Presence of Metabolic related arthritis (calcium crystal deposition, hemochromatosis, acromegaly)
* Arthritis related to trauma (major joint trauma, joint surgery)
* Presence of inflammatory disorders (rheumatoid arthritis, ankylosing spondylitis, septic arthritis)
* Previous surgical knee intervention
* Intraarticular injection of the knee in the previous 6 months.
* Presence of an unexpected traumatic episode in the affected knee (s) during the course of the study.
* Any contraindication for X ray or peripheral MRI study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Medial compartment knee cartilage thickness and volume | Baseline and after completion of 24 sessions
  A propietary software is been used to measure the cartilage thickness and volume of Magnetic Resonance Imaging obtained trough a coronal 3DGRE sequence. This measurement is been done by a trained physiatrist. The medial compartment is considered to be the primary outcome measure while the lateral compartment is considered as a secondary outcome.

SECONDARY OUTCOMES:
Western Ontario and McMaster Osteoarthritis Index Score (WOMAC) | Baseline and after completion of 24 sessions
  The Likert 3.1 version of the scale will be used.
Lower Extremity Functional Scale (LEFS) | Baseline and after competion of 24 sessions.
  The LEFS range from 0 (worst) to 80 (best)
6 minutes walk test | Baseline and after completion of 24 sessions
  The test will be conducted on a flat surface-rectangular hallway by instructing the participants to "Cover as much as distance as possible in a comfortable pace", the distance will be measured with a mechanical road distance measuring wheel (The Measure Meter ®, Truemeter 5500, UK), and the time was set using the timer function on an ipod touch. Standardized encouragement "you are doing fine, just keep going" will be given every minute.
Patient´s global assessment of disease severity (Likert scale 0- 5) | Baseline and after completion of 24 sessions
  Patients' perceptions of their disease severity was measured by the question "Considering all the ways knee osteoarthritis affects you, how would you rate your condition today?" and a Likert scale ( 1-very poor, 2- poor, 3- fair, 4-good, 5- very good).
Semi quantitative scoring of the knee joint | Baseline and after 24 sessions
  A semi quantitative score of MRI features related to the OA process (cartilage grade of injury, bone marrow edema, subchondral cyst) for each compartment (medial and lateral) along with independent scores of the medial meniscus, lateral meniscus, and joint effusion will be made by a trained radiologist
Pain at the end of the 6 minute walk test | Baseline and after 24 US sessions
  The level of pain at the end of the 6MT was recorded using a numeric pain scale ranging from 0 (no pain) to 10 (terrible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Norma J MacIntyre, PhD, Study Director — McMaster University; Julie Richardson, PhD, Study Chair — McMaster University; Karen Beattie, PhD, Study Chair — McMaster University; Adalberto Loyola-Sanchez, MD, Principal Investigator — McMaster University
Locations (1):
- School of Rehabilitation Science, Institute of Applied Health Sciences, McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Loyola-Sanchez A, Richardson J, Beattie KA, Otero-Fuentes C, Adachi JD, MacIntyre NJ. Effect of low-intensity pulsed ultrasound on the cartilage repair in people with mild to moderate knee osteoarthritis: a double-blinded, randomized, placebo-controlled pilot study. Arch Phys Med Rehabil. 2012 Jan;93(1):35-42. doi: 10.1016/j.apmr.2011.07.196. PMID 22200383